CLINICAL TRIAL: NCT01086397
Title: Distribution Of PCV13 Serotype Streptococcus Pneumoniae In Adults 50 Years And Older Presenting To Select US Hospitals With Radiographically-Confirmed Community-Acquired Pneumonia (CAP)
Brief Title: Epidemiologic Study Of The Distribution Of Vaccine-Type Streptococcus Pneumoniae Serotypes In Adults In The US With Community-Acquired Pneumonia
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 6115A1-4007; B1851032
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Pneumonia, Pneumococcal; Vaccines, Pneumococcal
Keywords: pneumococcal pneumonia; community-acquired pneumonia
MeSH Terms: conditions — Pneumonia, Pneumococcal; Community-Acquired Pneumonia

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine serum and potentially blood isolates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: Urine sample collection

INTERVENTIONS:
Procedure: Urine sample collection — All subjects have non-invasive urine sample collection performed

SUMMARY:
The main purpose of this study is to use an investigational urine assay to estimate the proportion of pneumonia in adults 50 years or older in different areas throughout the US that is caused by certain types of the bacteria Streptococcus pneumoniae (also called pneumococcus).

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and older.
* Presents to a study site with clinically suspected pneumonia.
* Has a radiographic finding that is consistent with pneumonia.
* Able and willing to provide urine.

Exclusion Criteria:

* Transfer to a study hospital after already being hospitalized for 48 hours or more at any other inpatient facility (such as community hospital).
* Hospital-acquired pneumonia (ie, pneumonia developing 48 hours after hospital admission).
* Previous enrollment in this study within the past 30 days.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 50 years and older presenting to Selected US Hospitals With Chest X-ray Confirmed Community-Acquired Pneumonia (CAP)
Sampling Method: Non-Probability Sample
Enrollment: 782 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have vaccine-type (VT), ie, PCV13, S. pneumoniae. | 6-12 months

SECONDARY OUTCOMES:
Proportion of subjects with VT-type pneumonia by previous healthcare facility exposure status will be described by site. | 6-12 months
Proportion of subjects with detection of S. pneumoniae by culture, BinaxNOW, and UAD assay will be summarized by method. | 6-12 months
Serotype distribution of S. pneumoniae cases by site and across all sites. | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - University of South Alabama Division of Clinical Research, Mobile, Alabama
  - Sharpe-Grossmont Hospital, La Mesa, California
  - Tampa General Hospital, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Detroit Receiving Hospital, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - eStudySite, Las Vegas, Nevada
  - Summa Infectious Diseases, Akron, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Sentara Norfolk General Hospital Cardiac Research 600 Gresh, Norfolk, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-4007&StudyName=Epidemiologic%20Study%20Of%20The%20Distribution%20Of%20Vaccine-Type%20Streptococcus%20Pneumoniae%20Serotypes%20In%20Adults%20In%20The%20US%20With%20Community-Acquired%20Pn